CLINICAL TRIAL: NCT06950346
Title: The Impact of TMS Ultrasound Curriculum on Learning Outcomes of PGY Emergency Physicians: A Retrospective Study
Brief Title: Online Ultrasound Curriculum on Learning Outcomes of Post-graduate Physicians
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202503116RINB
Record Dates: First submitted 2025-04-13; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Medical Education
Keywords: Medical education; Ultrasound; Online Training Management System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PGY trained with TMS ultrasound curriculum: PGY physicians trained with the TMS ultrasound curriculum participated in a structured, blended learning program that combined online modules with hands-on clinical training. The Training Management System (TMS) provided flexible, self-paced learning opportunities to reinforce foundational knowledge, while in-person sessions focused on skill application and image acquisition.

SUMMARY:
This single-center retrospective study evaluates the effectiveness of the Training Management System (TMS) ultrasound curriculum on the learning outcomes of PGY emergency physicians. By analyzing test scores and course participation data from 2018 to 2025, the study investigates whether blended learning improves PoCUS proficiency and explores its potential role in enhancing ultrasound education for junior physicians.

DETAILED DESCRIPTION:
Current point-of-care ultrasound education faces multiple challenges. Traditional teaching methods, such as didactic lectures and bedside one-on-one training, are constrained by time, clinical workload, and faculty availability, leading to inconsistent learning outcomes. Additionally, PGY physicians, due to their limited clinical experience, struggle to develop proficiency in ultrasound in a randomized learning environment. The quality of ultrasound image acquisition and diagnostic accuracy is also highly dependent on the operator's experience. In recent years, online learning platforms, such as the Training Management System, have been introduced to enhance learning flexibility. However, the long-term impact of such platforms on trainees' clinical application remains unclear. This study aims to evaluate the impact of the TMS ultrasound curriculum on the learning outcomes of PGY emergency physicians and explore the feasibility of a blended learning approach in improving ultrasound skill application. This single-center retrospective study analyzes test data from PGY trainees who participated in emergency PoCUS training between 2018 and 2025, including post-course test scores, objective structured clinical examination scores, and self-reported TMS course participation. The findings of this study may provide insights into the effectiveness of online and blended learning models in developing ultrasound proficiency among junior physicians and inform future medical education curriculum design.

ELIGIBILITY:
Inclusion Criteria:

1. PGY trainees who participated in the Department of Emergency Medicine ultrasound training program during the study period.
2. Trainees with complete course participation records and assessment results.

Exclusion Criteria:

1. Non-PGY participants (e.g., senior residents, attending physicians, medical students).
2. Incomplete assessment data that prevents a full evaluation of learning outcomes.
3. Any abnormal data not meeting study criteria (e.g., recording errors or duplicate entries).

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Postgraduate Year (PGY) trainees are newly graduated medical doctors undergoing structured clinical training as part of their early postgraduate education. In Taiwan, the PGY program is designed to enhance foundational clinical competencies through rotations across various medical specialties, including emergency medicine.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean Post-Course Test Score | From enrollment to the end of the test at 8 weeks
  Mean score of participants on the post-course knowledge test (range: 0-100 points; higher scores indicate better knowledge acquisition)
Mean OSCE Rating Score | From enrollment to completion of OSCE at 8 weeks.
  Mean score of participants on the Objective Structured Clinical Examination (OSCE) assessing ultrasound performance. The OSCE includes structured evaluation of the following domains:
  Image Acquisition Quality: Clarity and completeness of target anatomical structures (e.g., blood vessels, Morrison's pouch, spleno-renal recess, cul-de-sac).
  Diagnostic Accuracy: Ability to correctly interpret ultrasound findings and reach an appropriate clinical diagnosis.
  Scanning Technique and Efficiency: Smoothness, probe handling, and adherence to scanning protocols.
  Each domain is rated on a 10-point Likert scale (1 = Poor, 10 = Excellent), with higher scores indicating better clinical performance. The overall OSCE score is calculated as the mean of these domain scores.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Joji RM, Kumar AP, Almarabheh A, Dar FK, Deifalla AH, Tayem Y, Ismaeel AY, Bindayna K, Tabbara KS, Farid E, Shadab M, Al Mahmeed A, Shahid M. Perception of online and face to face microbiology laboratory sessions among medical students and faculty at Arabian Gulf University: a mixed method study. BMC Med Educ. 2022 May 30;22(1):411. doi: 10.1186/s12909-022-03346-2. PMID 35637505
- [Background] Harel-Sterling M. Can you teach a hands-on skill online? A scoping review of e-learning for point-of-care ultrasound in medical education. Can Med Educ J. 2023 Dec 30;14(6):66-77. doi: 10.36834/cmej.75272. eCollection 2023 Dec. PMID 38226294
- [Background] Lien WC, Chang CH, Chong KM, Wu MC, Wu CY, Wang HP. Clinical utilization of point-of-care ultrasound by junior emergency medicine residents. Med Ultrason. 2022 Aug 31;24(3):270-276. doi: 10.11152/mu-3425. Epub 2022 Jan 19. PMID 35045138